CLINICAL TRIAL: NCT06760390
Title: Cross-Sectional Analysis of Autonomic Differences in Heart Rate Variability Between Healthy Individuals and Subjects with Chronic Low Back Pain
Brief Title: Autonomic Differences in Heart Rate Variability Between Healthy and Chronic Low Back Pain Subjects
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Other Study IDs: 08
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Chronic Low Back Pain (CLBP); Heart Rate Variability; Autonomic Nervous System Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Subjects: This group includes adults aged 18-65 years without any chronic or acute pathology, no regular medication that could alter autonomic nervous system function, and no low back pain in the past six months.
- Chronic Low Back Pain Subjects: This group includes adults aged 18-65 years diagnosed with chronic low back pain lasting at least three months, with a minimum pain intensity of 3/10 on the Numerical Pain Rating Scale, and without uncontrolled neurological or cardiac disorders.

SUMMARY:
This study aims to evaluate the autonomic differences in heart rate variability (HRV) between healthy individuals and those with chronic low back pain. By analyzing HRV parameters, such as time-domain, frequency-domain, and non-linear metrics, this cross-sectional study seeks to explore the impact of chronic pain on the autonomic nervous system. The study will provide insights into parasympathetic and sympathetic modulation and its potential relationship with chronic pain symptoms. Participants include healthy adults and individuals with chronic low back pain aged 18-65.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years.

For the chronic low back pain group:

* Diagnosis of chronic low back pain lasting at least three months.
* A minimum pain intensity of 3/10 on the Numerical Pain Rating Scale (NPRS).

For the healthy group:

* Absence of any chronic or acute pathology.
* No regular medication that could alter autonomic nervous system function.
* No episodes of low back pain in the past six months.

Exclusion Criteria:

* Presence of uncontrolled neurological or cardiac disorders.
* Use of medications that could influence autonomic function or pain perception (e.g., opioids, antidepressants, benzodiazepines, anti-inflammatory drugs, beta-blockers) within two weeks prior to the study.
* Body Mass Index (BMI) equal to or greater than 30 kg/m².

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes two groups: one group of adults diagnosed with chronic low back pain, aged 18-65 years, and another group of healthy adults within the same age range. Participants were recruited from local community advertisements and hospital outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Root Mean Square of Successive Differences (rMSSD) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  This variable represents a time-domain measure of heart rate variability, reflecting parasympathetic nervous system activity and short-term variability in R-R intervals. It is calculated as the root mean square of differences between successive R-R intervals. rMSSD is an established metric to assess vagal modulation and is sensitive to changes in autonomic function.
SD1 (Short-Term Variability) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  A non-linear metric derived from the Poincaré plot of heart rate variability, indicating short-term variability in R-R intervals. It is closely associated with parasympathetic activity and vagal modulation.
SD2 (Long-Term Variability) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  A non-linear metric derived from the Poincaré plot, representing long-term variability in R-R intervals. SD2 is inversely related to sympathetic activity and reflects the balance between sympathetic and parasympathetic modulation.
Stress Score (SS) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  This variable is calculated as the reciprocal of SD2, multiplied by 1000. It reflects the level of sympathetic activation, where higher Stress Score values indicate increased stress and reduced parasympathetic activity.
Sympathetic/Parasympathetic Ratio (S/PS Ratio) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  This variable represents the ratio of Stress Score to SD1. It reflects the balance between sympathetic and parasympathetic modulation, with higher values indicating sympathetic dominance, commonly observed in chronic pain conditions.

SECONDARY OUTCOMES:
Mean Heart Rate (Mean HR) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  Represents the average heart rate (beats per minute) recorded during the data collection period. It serves as a general indicator of autonomic activity, providing insights into the balance between sympathetic and parasympathetic modulation.
Minimum Heart Rate (Min HR) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  Represents the lowest heart rate (beats per minute) recorded during the data collection period. This variable reflects periods of parasympathetic predominance and is useful for assessing vagal
Maximum Heart Rate (Max HR) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  Represents the highest heart rate (beats per minute) recorded during the data collection period. This variable reflects periods of sympathetic activation and provides insights into stress responses during the session.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D., Study Director — University of Extremadura
Locations (1):
- Universidad de Extremadura, Badajoz, Badajoz, Spain